CLINICAL TRIAL: NCT02727257
Title: The Effect of a Motor-cognitive Rehabilitation on Attention in Parkinsonian Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rehabilitation and RT in PD
Record Dates: First submitted 2016-03-06; First posted 2016-04-04 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; rehabilitation; attention; executive functions
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIRT (Experimental): MIRT consists of a 4-week physical therapy that entails four daily sessions, five days a week, in a hospital setting. The first session comprise cardiovascular warm-up activities, relaxation, muscle-stretching, exercises to improve the range of motion of spinal, pelvic and scapular joints, exercises to improve the functionality of the abdominal muscles, and postural changes in the supine position. The second session includes aerobic exercises to improve balance and gait using a stabilometric platform, treadmill plus, crossover and cycloergometer. All the exercises are aerobic. The third is a session of occupational therapy to improve autonomy in day living activities. The last session includes one hour of speech therapy.
  Interventions: Procedure: MIRT
- healthy controls (No Intervention): we assessed the attentive Reaction Times in healthy controls, that don't receive rehabilitative treatment

INTERVENTIONS:
Procedure: MIRT — MIRT consists of a 4-week physical therapy that entails four daily sessions, five days a week, in a hospital setting. The duration of each session, including recovery periods, is about one hour. The first session comprise cardiovascular warm-up activities, relaxation, muscle-stretching, exercises to improve the range of motion of spinal, pelvic and scapular joints, exercises to improve the functionality of the abdominal muscles, and postural changes in the supine position. The second session includes aerobic exercises to improve balance and gait using a stabilometric platform, treadmill plus, crossover and cycloergometer. The third is a session of occupational therapy to improve autonomy in day living activities. The last session includes one hour of speech therapy.
  Arms: MIRT

SUMMARY:
In this study the Investigators explore two questions: if the attentive reaction times differs in parkinsonian patients from health controls and if an intensive, focused and aerobic rehabilitation program (Multidisciplinary Intensive Rehabilitation Treatment - MIRT) tailored mainly for motor problems, could have a specific positive effect on multiple choices Reaction Times (RTs) as an indirect marker for an effect on attentional-executive frontal circuits. The hypothesis is that the MIRT could have a positive effect on the top-down control mechanisms, since the continuous feedback given by physiotherapist during exercises and the use of cues and devices (such as treadmill plus and stabilometric platform), stimulate the selective attention processes that enable goal-directed, internally-driven decision, helping the patients to overcome externally-driven decision based on stimulus salience and novelty

DETAILED DESCRIPTION:
Objective: To evaluate the attentive performances in Parkinsonians in comparison with healthy controls and the effect of motor-cognitive rehabilitation program on attention.

Methods: 103 Parkinsonians (stage 2,5-3 H&Y) hospitalized for a 4-week Multidisciplinary Intensive Rehabilitation Treatment and 34 healthy controls were enrolled. All subjects underwent three different attentive tasks: visual reaction times, auditory reaction times and multiple choices reaction times tasks. To evaluate the effect of rehabilitation on attention, patients performed the same battery at discharge. To investigate the effects of MIRT on motor functions and quality of life we also assessed UPDRS III, Timed Up and Go test and Parkinson's Disease Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* stage 2.5-3 according to the Hoehn & Yahr scale
* pharmacological treatment for the last 8 weeks and during the hospitalization
* Mini Mental State Examination (MMSE) ≥ 24

Exclusion Criteria:

* any focal brain lesion detected in brain imaging studies (Computed Tomography or Magnetic Resonance Imaging) performed in the previous twelve months
* disabling drug-induced dyskinesias
* disturbing resting and/or action tremor, corresponding to scores 2 to 4 in the specific items of Unified Parkinson's Disease Rating Scale section 3 (UPDRS III)
* behavioral disturbances (evaluated with Neuropsychiatric Inventory)
* visual and auditory dysfunctions according to the general clinical evaluation and medical history

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Multiple Choice Reaction Time task | 4 weeks
  The task consisted of 40 trials. The target was a number (1, 2, 3) whose presentation, on the centre of the screen, was randomized. Each number was associated to a different response buttons . In each single trial subjects had to press as quickly as possible the response button associated with the number that appeared on the screen. We evaluated the accuracy of response and recorded the time between the appearance of target and the subject's response.

SECONDARY OUTCOMES:
Simple Choice Reaction Time task | 4 weeks
  The task consisted of 40 trials. In each single trial, the subjects had to press the response button as quickly as possible when a red circle appeared on the screen. The appearance of targets was mixed to a variable number of distractors consisting in single green circles. Targets and distractors could appear in different positions of the screen at irregular intervals (1-3 seconds). Distractors remained on the screen for 500 ms, while the target disappeared with the subject's response. We evaluated the accuracy of response and recorded the time between the appearance of target and the subject's response.

OTHER OUTCOMES:
Auditory Reaction Time task | 4 weeks
  The task consisted of 40 trials. In each single trial the subjects had to press a response button as quickly as possible at the presentation of the target that consisted of an acoustic stimulus (intensity of 94 dbA) presented at irregular intervals (1-3 seconds). The stimulus ended after the subject's response. The times between the presentation of the target and the subject's response were recorded.
Visual Reaction Time task | 4 weeks
  The task consisted of 40 trials. In each single trial, the subjects had to press a response button as quickly as possible at the appearance of the target that disappeared after the subject's response. Target was a red circle that appeared on the centre of screen at irregular intervals (1-3 seconds). The times between the appearance of the target and the subject's response were recorded.
Unified Parkinson's disease Rating Scale | 4 weeks
Parkinson Disease Questionnaire - 39 | 4 weeks
Timed Up and Go Test | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital - Gravedona ed Uniti (CO, Italy)
Locations (1):
- Department of Parkinson's Disease and Brain Injury Rehabilitation, of the 'Moriggia-Pelascini' Hospital, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No